CLINICAL TRIAL: NCT00681083
Title: Titrations Pressures in Sleep Apnea Patients Using ThermoSmart® Versus Conventional Humidification
Brief Title: Titration Pressures in Sleep Apnea Patients Using ThermoSmart® Versus Conventional Humidification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Collaborators: Sleep Disorder Centers Institute for Clinical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FPHC SDC 2008
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2019-06-12 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-05

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea; Humidification; Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Heated breathing tube
  Interventions: Device: Heated breathing tube (CPAP with ThermoSmart)
- 2 (Active Comparator): Non heated breathing tube
  Interventions: Device: Non heated breathing tube (CPAP with conventional humidification)

INTERVENTIONS:
Device: Heated breathing tube (CPAP with ThermoSmart) — CPAP with ThermoSmart - heated passover humidifier, with heated breathing tube
  Other Names: ThermoSmart
  Arms: 1
Device: Non heated breathing tube (CPAP with conventional humidification) — CPAP with conventional humidification - heated passover humidifier, no heated breathing tube
  Other Names: Conventional humidification
  Arms: 2

SUMMARY:
Patients who have Obstructive Sleep Apnea (OSA) may have different Continuous Positive Airway Pressure (CPAP)when titrated with different levels of humidification. It is hypothesised that patients with ThermoSmart® technology (heated breathing tube technology) will have lower titrated pressures than those who are titrated using conventional humidification (non heated breathing tube).

DETAILED DESCRIPTION:
Debate is present concerning the optimal level of humidification for obstructive sleep apnea (OSA) patients who need continuous positive airway pressure (CPAP) therapy. Recent evidence has shown that using a heated breathing tube to increase the amount of humidification that can be delivered has decreased patient side effects, increased subjective sleep quality and decreased subjective symptom scores. Anecdotal evidence exists, in the form of clinical observation, when ThermoSmart® technology is utilized during CPAP titration, patients laboratory titrated pressure may in fact prove to be lower. The possibility exists, on a titration night, patients potentially may experience an adverse response to the positive airway pressure which manifests as increased airway resistance and inflammation necessitating higher CPAP pressures to overcome upper airway resistance and flow limitation. Therefore, we hypothesize the delivery of higher levels of humidity might reduce the nasal airway resistance during the titration night, reducing the overall positive airway pressure requirements. The goal is to investigate this phenomenon to find if a reduction in pressure is necessary and if so to what degree. Patients who are titrated on Continuous Positive Airway Pressure devices with ThermoSmart® technology will have lower titrated pressures than those who are titrated using conventional humidification.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female patients over the age of 18
* Apnea Hypopnea Index (AHI) ≥15
* Patients must have at least 5 hours sleep time on each titration night
* Stable medications for 2 weeks prior to entry to the study and for study inclusion duration including sleep aids

Exclusion Criteria:

* Receiving or requiring bi-level ventilation
* Use of a full face interface or chin strap
* Previous UPPP surgery or palatal reconstruction
* Recent angina symptoms within 2 weeks of entry
* CHF with EF < 40%
* Obesity Hypoventilation Syndrome
* Cheyne Stokes respiration
* > 50% Central apneas recorded on diagnostic polysomnogram
* Supplemental oxygen use
* Use of narcotic pain medication
* Hypoxemia as determined by room air pulse oxymetry of less than 89% on room air at rest awake
* Inability to tolerate positive pressure therapy
* Split Night Evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Lewis, M.D., Principal Investigator — Sleep Disorder Centers Institute for Clinical Research
Locations (2):
- United States (2):
  - Sleep Center of Tulsa - Midtown, Tulsa, Oklahoma
  - Sleep Center of Tulsa - South, Tulsa, Oklahoma

REFERENCES:
- See also: Fisher & Paykel Healthcare — http://www.fphcare.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Heated Breathing Tube: Heated breathing tube (CPAP with ThermoSmart): CPAP with ThermoSmart - heated passover humidifier, with heated breathing tube
- Non Heated Breathing Tube: Non heated breathing tube (CPAP with conventional humidification): CPAP with conventional humidification - heated passover humidifier, no heated breathing tube
Period: Night 1
Arm/Group | Heated Breathing Tube | Non Heated Breathing Tube
Started | 13 (26 participants were initially consented (this is the total for the study).) | 13 (26 participants were initially consented (this is the total for the study).)
Completed | 10 (20 in total completed study. 10 randomized to arm 1 and arm 2 then crossed over to other arm.) | 10 (20 in total completed study. 10 randomized to arm 1 and arm 2 then crossed over to other arm.)
Not Completed | 3 | 3
Period: Night 2 (Crossover of Night 1)
Arm/Group | Heated Breathing Tube | Non Heated Breathing Tube
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All Study participants. Note: participants took part in both arms as it was a cross over trial
Arm/Group | All Study Participants
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 48.35 [21 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Titration Pressures After Treatment Nights
Description: Each night, the participant underwent a CPAP titration to determine their therapeutic pressure. During a titration, a sleep technician manually adjusts the participants pressure to determine which pressure is best for that individual in reducing their Apnea Hypopnea Index (AHI) which is the measure of Obstructive Sleep Apnea (OSA) severity. Titration pressures for each group were compared to see if there was any impact of having a heated breathing tube versus a non heated breathing tube on titration pressure.
Time Frame: End of titration night
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Heated Breathing Tube | Non Heated Breathing Tube
Number analyzed (Participants) | 20 | 20
cmH20 | 9.8 (1.89) | 10.9 (1.98)

2. Secondary Outcome: Relationship Between the Intervention (Heated Breathing Tube vs Non Heated Breathing Tube) and Total Sleep Time
Description: A correlation table was computed to explore the relationship between the intervention (heated breathing tube vs no heated breathing tube) and total sleep time. This relationship was calculated for each arm and reported by a Correlation Coefficient (r score). The r score represents the strength and direction of a relationship between two variables. The value of r is always between -1 and +1. Therefore, an r score of -1 indicates a perfect negative relationship between the intervention and total sleep time. An r score of -.50 indicates a moderate negative relationship between the intervention and total sleep time. An r score of 0 indicates no relationship between the intervention and total sleep time. An r score of +.50 indicates a moderate positive relationship between the intervention and total sleep time. An r score of +1 indicates a perfect positive relationship between the intervention and total sleep time.
Time Frame: End of titration night
Measure: Number; unit: r score
Arm/Group | Heated Breathing Tube | Non Heated Breathing Tube
Number analyzed (Participants) | 20 | 20
r score | .535 | .058

ADVERSE EVENTS:
Arm/Group | Heated Breathing Tube | Non Heated Breathing Tube
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other